CLINICAL TRIAL: NCT02099227
Title: Comparative Effectiveness of Emergency Ultrasound Guided Management of Pediatric Soft Tissue Infections
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American College of Emergency Physicians (Other); Newark Beth Israel Medical Center (Other); Baylor College of Medicine (Other); UCSF Benioff Children's Hospital Oakland (Other); Maimonides Medical Center (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: AHC IRB 5577
Record Dates: First submitted 2014-03-26; First posted 2014-03-28 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2016-09

CONDITIONS: Soft Tissue Infection
Keywords: pediatric; soft tissue infections; ultrasonography; effectiveness
MeSH Terms: conditions — Soft Tissue Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ultrasound: those who received point-of-care ultrasound as part of their emergency department evaluation/ treatment for suspected soft tissue infections
- No Ultrasound: those who did not receive point-of-care ultrasound as part of their emergency department evaluation/ treatment for suspected soft tissue infections

SUMMARY:
To examine the effect of Point-of-Care Ultrasound (POCUS) management guidance on pediatric skin and soft tissue infections treatment failure rate, as well as emergency department process outcome.

ELIGIBILITY:
Inclusion Criteria:

* history and examination findings consistent with possible abscess or cellulitis per the treating clinician.
* minimal lesion diameter for inclusion is 1cm.

Exclusion Criteria:

* suspected soft tissue infections involving or near mucosal membranes (e.g. perirectal, peritonsillar, vulvovaginal areas)
* facial lesions
* paronychia or felon
* parent or patient refusal of consent
* unsuitable subjects deemed by treating clinicians.

Ages: 6 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children presenting to participating pediatric emergency departments
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
treatment failure rate | 7-10days
  unscheduled return visits need for subsequent procedural intervention need for subsequent admission change in therapy

SECONDARY OUTCOMES:
emergency department process outcome | 7-10days
  emergency department (ED) length of stay, need for ED procedural sedation use of alternative imaging in ED

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Lam, MD, Principal Investigator — advocate christ medical center
Locations (1):
- Advocate Christ Medical Center, Oak Lawn, Illinois, United States